CLINICAL TRIAL: NCT01267786
Title: The Effect of Volatile Anesthetics Sevoflurane and Desflurane on Liver, Renal and Cardiovascular Systems During Liver Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieio Hospital (Other)
Responsible Party: G.P. Fragulidis MD, Ass. Prof. Surgery, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AnesthSurg1
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Apoptosis; Liver Surgery
Keywords: Oxidotic stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane (Active Comparator): 1MAC intraoperatively
  Interventions: Procedure: Liver surgery
- desflurane (Active Comparator): 1 MAC intraoperatively
  Interventions: Procedure: Liver surgery

INTERVENTIONS:
Procedure: Liver surgery — hepatectomy

SUMMARY:
The aim of the study is to investigate the effect of sevoflurane and desflurane on hepatic function after ischemic/reperfusion injury and the sequence influence on renal and cardiovascular systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver surgery

Exclusion Criteria:

* ASA IV, Cardiovascular diseases

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Oxidotic stress after hepatectomy. | 5 d postop.
  Perioperative liver and renal biopsies and follow up with liver renal function tests plus intraoperative and postoperative cardiovascular monitoring

SECONDARY OUTCOMES:
Liver and renal dysfunction | 5 d
  liver and renal impairment due to ischemic injury

CONTACTS AND LOCATIONS:
Overall Officials: Georgios P Fragulidis, MD, Principal Investigator — Areataieio Hospital
Locations (1):
- Aretaieio Hospital, Athens, Attica, Greece